CLINICAL TRIAL: NCT07311616
Title: A Study on the Effectiveness of Preventive Extensive Release of the Rotator Interval and Joint Capsule to Reduce Postoperative Stiffness in Arthroscopic Rotator Cuff Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MR-11-25-079098
Record Dates: First submitted 2025-11-30; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Supraspinatus Tear
Keywords: Rotator cuff repair; Postoperative stiffness; Joint capsule release; Randomized controlled trial; Range of motion of the shoulder joint
MeSH Terms: interventions — Joint Capsule Release

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group underwent arthroscopic rotator cuff repair combined with preventive extensive shoulder release and capsular release simultaneously.
  Interventions: Procedure: Prophylactic extensive shoulder release and capsular release; Procedure: Arthroscopic rotator cuff repair
- Control Group (Other): The control group only received arthroscopic rotator cuff repair surgery.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Prophylactic extensive shoulder release and capsular release — Before rotator cuff repair, extensive release of the rotator cuff space is performed first, as well as comprehensive release of the middle glenohumeral ligament, inferior glenohumeral ligament, coracohumeral ligament, the area around the subscapularis tendon, the subacromial capsule, and the anterior and posterior inferior joint capsules.
  Arms: Experimental Group
Procedure: Arthroscopic rotator cuff repair — Arthroscopic rotator cuff repair surgery

SUMMARY:
The incidence of rotator cuff injuries is high, especially among the elderly. With the aging of the population, the number of surgical patients has increased significantly. However, in the early stage after arthroscopic rotator cuff repair, a considerable proportion of patients are troubled by shoulder joint stiffness, which greatly affects the quality of life and satisfaction of patients after the operation. Despite this, there is still a lack of clear evidence-based medical evidence regarding whether preventive extensive shoulder release and joint capsule release during arthroscopic rotator cuff repair can effectively prevent or alleviate postoperative shoulder stiffness. To clarify this clinical issue, this project intends to conduct a single-blind randomized controlled trial (RCT). Before the operation, patients will be randomly divided into two groups under blinding conditions: the experimental group will receive arthroscopic rotator cuff repair surgery along with preventive extensive shoulder joint release and joint capsule release, while the control group will only receive arthroscopic rotator cuff repair surgery. After the operation, the investigators will conduct follow-up visits for 3 months, 6 months and 12 months for the two groups of patients, and perform magnetic resonance imaging (MRI) at the 12th month to assess the healing of the rotator cuff tendons. ASES score, Constant-Murley score, Visual Analogue Scale (VAS) pain score and active range (ROM) assessment were conducted before the operation and at the follow-up at 3 months, 6 months and 12 months after the operation. The occurrence of postoperative complications of the patients was counted at the last follow-up. Through this study, the investigators expect to provide scientific and effective guidance for the prevention of postoperative adhesions of the shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

1. Medium to small-sized (tear size <3 cm) full-thickness supraspinatus muscle tears
2. There was no shoulder joint stiffness before the operation. The range of motion of the joint was at least 160° for passive forward flexion under ROM anesthesia, 60° for external rotation when abduction was 0°, and equal to or greater than 60° for passive internal rotation at the level of the 10th thoracic vertebra
3. About to undergo ARCR
4. No history of trauma
5. Patient consent to participate

Exclusion Criteria:

1. There was a history of previous surgery on the ipsilateral shoulder
2. Other injuries or lesions of the ipsilateral shoulder (such as glenohumeral arthritis, combined acromioclavicular joint dislocation, brachial plexus injury, etc.)
3. It can not be completely repaired or even repaired during operation
4. Have uncontrolled epilepsy or psychological illness
5. Patients who were assessed as not suitable for inclusion in the study group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Daily Functional Evaluation Measured By American Shoulder and Elbow Surgeons Score (ASES Questionnaire) | At baseline and at 3, 6 and 12 months after the operation.
  This outcome measure will be assessed using the American Shoulder and Elbow Surgeons Score (ASES), a disease-specific patient-reported outcome questionnaire. The scale consists of two key dimensions: pain (50 points, measured by Visual Analog Scale) and daily living functions (50 points, evaluating 10 activities including dressing, combing hair, and using the toilet). The total score ranges from 0 to 100, with higher scores indicating better shoulder function and less pain.

SECONDARY OUTCOMES:
Shoulder Function Measured By Constant-Murley Score | At baseline and at 3, 6 and 12 months after the operation.
  The Constant - Murley Score is a validated scale developed in 1986 for evaluating shoulder joint function, consisting of four assessment dimensions. It includes pain level (15 points), daily living activities (20 points), shoulder range of motion (40 points), and muscle strength (25 points), with a total score of 0 - 100. A higher score indicates better shoulder joint function. The subjective parts (pain and daily living activities) are completed by subjects themselves, while the objective parts (range of motion and muscle strength) are evaluated and recorded by researchers.
Patient-Reported Shoulder Pain Intensity Measured by Visual Analogue Scale (0-10 Scale) | At Basline, 1 day after the operation, and 3, 6, and 12 months after the operation
  This outcome measure evaluates the intensity of shoulder pain in patients with supraspinatus muscle tear. A 100mmVAS ruler is used as the measurement tool (0mm= no pain, 100mm= extreme pain) to measure the intensity of shoulder pain in participants at baseline, 1 day after operation, 3 months, 6 months and 12 months of follow-up. Record the changes in VAS scores from baseline to each time point to reflect the intervention effect.The Visual Analogue Scale ranges from a minimum of 0 to a maximum of 10, and the higher the score, the worse the result.
Range of Motion (ROM) | At baseline and at 3, 6, and 12 months after operation
  Postural photos were taken to measure the Angle of joint movement
Rate of Postoperative Complications | At 6 weeks, 3 months, 6 months and 12 months after the operation.
  Inquire about the medical history to identify postoperative complications in paticipants.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified individual participant data, study protocols, statistical analysis plans, and summaries of clinical study reports. These data include all variables analyzed in the primary and secondary outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available beginning 6 months after the publication of the primary study results and will remain accessible for at least 3 years.